CLINICAL TRIAL: NCT04266496
Title: Discovering the Effect of Venous Insufficiency on Nocturia: a Prospective, Controlled Trail
Brief Title: Discovering the Effect of Venous Insufficiency on Nocturia
Acronym: DEVINe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BC-6121
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Nocturia; Venous Insufficiency of Leg; Fluid Overload
MeSH Terms: conditions — Nocturia; Edema | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- <2 nocturnal voids (Other): All interventions in this group are done twice: Once before surgical intervention, and once 2 months after surgical intervention
  * Complete a 3 day Frequency Volume chart
  * Questionnaires: ICIG FLUTS/MLUTS, PSQI and CIVIQ2
  Interventions: Other: Questionnaires; Diagnostic Test: Frequency Volume Chart
- => 2 nocturnal voids (Other): All interventions in this group are done twice: Once before surgical intervention, and once 2 months after surgical intervention
  * Complete a 3 day Frequency Volume chart and collection of the urine of the last day and night to complete osmolality and sodium testing.
  * Measuring the circumference off the lower limbs just after awakining and before falling asleep
  * Questionnaires: ICIG FLUTS/MLUTS, PSQI and CIVIQ2
  Interventions: Other: Questionnaires; Diagnostic Test: Frequency Volume Chart; Diagnostic Test: Collect urine during 1 day; Diagnostic Test: Blood sample; Diagnostic Test: Measurement of the circumference of the lower legs

INTERVENTIONS:
Other: Questionnaires — ICIQ FLUTS (women) or MLUTS (mannen) CIVIQ 2 PSQI
Diagnostic Test: Frequency Volume Chart — Collect a frequency volume chart for 3 days: measure the amount of voids and volume urinated.
Diagnostic Test: Collect urine during 1 day — Volunteers are asked to collected their urine during the last day of the frequency volume chart. Volunteers get 2 jars: One for collection during the day, and 1 for overnight collection of urine. Osmolality and sodium of urine is tested
  Arms: => 2 nocturnal voids
Diagnostic Test: Blood sample — Blood collection to measure plasma sodium and osmolality.
  Arms: => 2 nocturnal voids
Diagnostic Test: Measurement of the circumference of the lower legs — Circumference of the lower legs wil be measured twice:
  * After awakening, when still laying dowing in bed
  * Before goin to sleep
  Circumference should be measured 2 cm above the medial malleolus
  Arms: => 2 nocturnal voids

SUMMARY:
With this prospective controlled trial, we hope to obtain more information about the coexistence between venous insufficiency and nocturia.

In our opinion, venous insufficiency (CEAP 2-3a) leads to an increase in fluid accumulation in the lower limbs due to moving around all day. When laying down during nighttime, this fluid is reabsorbed into the systimic fluid pool, leading to an increase in diuresis and thus an increase in nocturnal voiding. Aim of this study is observe difference in nocturnal frequency and urine production before and after surgical treatment of venous insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* CEAP 2 till 4A

Exclusion Criteria:

* BMI higher than 30
* Previous surgery due to venous insufficiency at the lower limbs
* Cronic edema (Cronic heart failure, liver cirrosis, nefrotic syndrome)
* Pregnant patient
* Patients on the following medication: Calcium-antagonists, lithium, NSAID's or corticosteroids, glitazones, insuline, diuretics, sartans, ACE-inhibitors, desmopressine,

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Change of micturition frequency | 2 months after surgery
  Change of the micturition frequency with 1 void

SECONDARY OUTCOMES:
Change in nocturnal diuresis | 2 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Karel Everaert, MD PhD, Principal Investigator — UZ Ghent
Locations (1):
- Department of urology, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided